CLINICAL TRIAL: NCT04367506
Title: Pilot Testing a Digital Intervention to Improve Smoking Cessation in Persons With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Sheppard Pratt Health System (Other); Truth Initiative (Other)
Responsible Party: Principal Investigator, Melanie E Bennett, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH120142 (NIH)
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: This project has three phases. Phase 1: Adapt BecomeAnEX, conduct usability testing (n=10), and train digital coaches. Phase 2: Conduct a 1-arm pilot trial of the adapted BecomeAnEX (n=20). Phase 3: Conduct a pilot randomized controlled trial (n=90) to examine indicators of feasibility, acceptability, target mechanisms, and preliminary efficacy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BecomeAnEX (Experimental): Participants will have three individual meetings with a research staff person while they are in the hospital. At these meetings participants will answer questions about their smoking and interest in quitting, learn about BecomeAnEx, and register with the BecomeAnEx program so that they can use it when you leave the hospital. Participants will be given two weeks of nicotine replacement therapy when they leave the hospital. Participants will be asked to use BecomeAnEx as much as they want when they leave the hospital.
  Interventions: Behavioral: BecomeAnEX; Behavioral: Usual Care
- Usual Care (Active Comparator): Brief individual counseling, NRT during the hospital stay and a prescription for NRT at discharge (consistent with standard hospital procedures), and referral to the MD quitline.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: BecomeAnEX — This research study is focused on a smoking cessation program called BecomeAnEx. We are studying how to adapt BecomeAnEx for people with a mental health disorder who want to reduce or quit their tobacco smoking. BecomeAnEx includes a website that provides education about smoking and quitting. It also has a text messaging program that delivers personalized information. Persons in the program have access to real-time digital coaching with a remote coach who has experience helping people quit smoking. In addition, the program has an on-line community of current and former smokers that can provide support and encouragement.
  Arms: BecomeAnEX
Behavioral: Usual Care — Usual care represents what hospitalized psychiatric patients normally receive in terms of smoking cessation: brief individual counseling, NRT during the hospital stay and a prescription for NRT at discharge (consistent with standard hospital procedures), and referral to the MD quitline.

SUMMARY:
All patients with serious mental illness are abstinent while in the hospital for a psychiatric admission yet almost all return to smoking after discharge. The investigators propose to adapt a digital intervention both to the needs of SMI smokers and to being introduced in the inpatient psychiatric setting through a collaboration between experts in SMI and the Truth Initiative, a pre-eminent tobacco control organization. The investigators believe this will bridge the inpatient to outpatient gap in cessation services and will help people remain abstinent following hospital discharge.

DETAILED DESCRIPTION:
Persons with serious mental illness (SMI) die on average 10-15 years earlier than those in the general population. Smoking is the strongest risk factor for their elevated mortality. Helping SMI smokers to quit is an urgent and unmet need. The hospital is an optimal setting to provide smoking cessation services. Hospital admissions for SMI are common with more than 1.2 million inpatient stays for schizophrenia and mood disorders per year in the US. Hospitalized patients experience required abstinence, are available for counseling, and can try cessation medications in a supportive setting. The challenge is how to engage SMI patients in cessation services post-discharge. An easy-to-access digital intervention is a scalable and sustainable way to bridge the inpatient-to-outpatient gap and to promote sustained abstinence. Digital interventions can deliver all elements of cessation treatment and yield quit rates comparable to face to face and telephonic interventions. SMI patients use and benefit from technology-based interventions but currently there is no digital smoking cessation program addressing their needs. This R34 application will adapt a proven digital intervention, BecomeAnEX (EX), developed and run by Truth Initiative for over 10 years. Its core components are real-time one on one coaching via live chat, nicotine replacement therapy decision support and delivery, personalized quit plans, a large online social network for peer support, a robust and fully integrated text message program, and tailored email messaging. Adaptation will ensure that EX addresses the specific challenges of SMI smokers and is in line with principles of mental health recovery. In Aim 1 the investigators will develop and obtain preliminary feedback about EX-SMI, a version of EX adapted for SMI patients. A priori target mechanisms are motivation, abstinence self-efficacy, and cravings. In Aim 2 the investigators will conduct a one-arm pilot trial and obtain feedback from 20 SMI smokers recruited during psychiatric hospitalization and followed up at 2-weeks and 1-month post-discharge. Feasibility and acceptability will be assessed via participant feedback regarding their intervention experience, changes in motivation, self-efficacy and cravings, and automated tracking data on EX-SMI use post-discharge. In Aim 3, 90 SMI smokers recruited during psychiatric hospitalization will be randomized to usual care or to a revised version of EX-SMI and followed for 3 months after the hospital stay. The investigators will compare the feasibility/acceptability of EX-SMI, measure intervention impact on target mechanisms, and obtain initial estimates of efficacy on 7-day point prevalence abstinence. This pilot work directly addresses priorities of this RFA in refining and optimizing an efficacious intervention for a new target population. Ultimately, this program of research could have a powerful public health impact by increasing smoking cessation among persons with SMI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Diagnosis of serious mental illness (schizophrenia, schizoaffective disorder, bipolar disorder, or major depression)
* Current smoker [prior to admission, smoked at least one cigarette or small cigar per day in the past month (unless restricted, e.g. due to ER/hospital visit) and smoked at least 100 cigarettes lifetime]
* Interested in remaining quit after hospital discharge or quitting within the following 30 days
* Expected Internet use at least 3 times/week post-discharge and ownership of mobile device with text messaging plan post-discharge.
* Discharge destination within 1-hour of SPH given that Aim 3 involves biochemical verification (carbon monoxide testing).
* Reading competence as demonstrated by a score of >= 37 on the Word Reading subtest of the Wide Range Achievement Test - 4th Edition (WRAT-4)168 to ensure the ability to engage in the intervention.

Exclusion Criteria:

* Intellectual disability (DSM5 317, 318), traumatic brain injury, or deafness.
* Homeless prior to admission or anticipated to be homeless at discharge.
* Discharge to a residential setting where smoking is prohibited.
* Medical condition for which the use of nicotine replacement therapy (NRT) is contraindicated including pregnant, planning to become pregnant, or breastfeeding; within 4 weeks post myocardial infarction; severe arrhythmia, severe angina pectoris; peptic ulcer; severe renal failure; poorly controlled insulin-dependent diabetes; severely uncontrolled hypertension; peripheral vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 1 month
  Self-report 7-day point prevalence abstinence
Craving | 1 month
  Tobacco Cravings Questionnaire
Self-efficacy | 1 month
  Smoking Situations Confidence Questionnaire
Motivation to remain abstinent | 1 month
  Abstinence-Related Motivational Engagement Scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Melanie Bennett, Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland